CLINICAL TRIAL: NCT01978574
Title: A Randomized Controlled Trial of Intellectual Enrichment to Build Cognitive Reserve in Multiple Sclerosis
Brief Title: Intellectual Enrichment to Build Cognitive Reserve in MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NMSS-PP1854
Record Dates: First submitted 2013-10-31; First posted 2013-11-07 (Estimated); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Cognitive Impairment in Multiple Sclerosis
Keywords: Cognitive reserve; intellectual enrichment

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Documentary videos (Active Comparator): In the placebo control condition, participants watch daily videos.
  Interventions: Behavioral: Intellectual Enrichment documentary videos
- Intellectual Enrichment (Experimental): Daily activities that encourage intellectual enrichment, including games, reading/writing, and hobby activities.
  Interventions: Behavioral: Intellectual Enrichment daily activities

INTERVENTIONS:
Behavioral: Intellectual Enrichment daily activities — A daily program of intellectually enriching, iPad/tablet-based activities: games, reading/writing, hobby activities, or a documentary video (control).
  Arms: Intellectual Enrichment
Behavioral: Intellectual Enrichment documentary videos — Participants watch daily documentary videos.
  Other Names: Placebo control condition
  Arms: Documentary videos

SUMMARY:
Cognitive problems are a primary concern for people with multiple sclerosis. In many cases, people with MS report these issues to be more debilitating than the motor symptoms that are targeted by most treatment strategies. For people with MS, impaired memory and thinking skills can interfere with the ability to function efficiently in multiple professional and personal roles. Finding ways to decrease, slow, or reverse declines in memory and thinking skills is a vitally important research priority. We now know that engaging in intellectually enriching activities helps protect against the negative impact of MS disease-related declines in memory and thinking. Such activities contribute to something called 'cognitive reserve,' which serves as a protection against disease-related declines in memory and thinking. Thus far, no one has created a treatment that aims to provide a concentrated 'dose' of intellectual enrichment to build cognitive reserve. The present intervention aims to do precisely this. Here, we have developed a program of enriching activities that are delivered via a personal iPad. This allows for a 12-week 'treatment' that is entirely home-based, while also providing close personal contact between participants and our study personnel, who will communicate daily via emails. Week by week, participants choose from a menu of intellectually enriching activities such that their treatment is dynamic and customizable to fit their interests. The intervention is designed to be fun, as we hope the activities will be incorporated into people's lives beyond the period of the study itself. Given what we already know about the striking benefits of cognitive reserve to protect against disease-related declines in cognitive functioning, we expect to show that treatment with a daily, intense, intellectually enriching schedule of activities results in improved thinking and memory for people with MS. We will also investigate the positive impact of our treatment on the brains of people with MS through brain scans. We expect to see evidence for a shift toward more efficient processing in the brain, changes that translate to improved memory and thinking skills.

ELIGIBILITY:
Inclusion Criteria:

* age 25-65
* MS duration >5 years
* read and speak English fluently

Exclusion Criteria:

* currently experiencing an MS exacerbation
* MS exacerbation within 6 weeks of study start
* left handed
* non-MRI compatible: metal in body, claustrophobic
* history of neurological disorder other than MS
* history of head injury
* history of schizophrenia or bipolar disorder
* pregnant
* currently taking steroids, benzodiazepines, and/or neuroleptics
* do not speak English as primary language

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-06-01 (Actual); Primary Completion 2014-06-01 (Actual); Study Completion 2014-06-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Hopkins Verbal Learning Test and Brief Visuospatial Memory Test, Total Learning and Delayed Recall | Baseline and 13 weeks

SECONDARY OUTCOMES:
Change from Baseline in Beck Depression Inventory | Baseline and 13 weeks

OTHER OUTCOMES:
Change from Baseline in fMRI task-related BOLD activation pattern | Baseline and 13 weeks
  A neural pattern of fMRI BOLD activation indicating cerebral efficiency will be assessed at baseline and follow-up.
Change from Baseline in fMRI-derived functional connectivity | Baseline and 13 weeks
  A neural pattern of fMRI functional connectivity will be assessed at baseline and follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria M Leavitt, PhD, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States